CLINICAL TRIAL: NCT03591003
Title: "Persistence of Neutralizing Antibodies After Immunization Against Yellow Fever (YF) in HIV-infected Patients: a Multicenter Study"
Brief Title: "Persistence of Neutralizing Antibodies Against Yellow Fever (YF) in HIV-infected Patients"
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Charlotte Martin, Infectious Diseases Senior Resident, Centre Hospitalier Universitaire Saint Pierre
Other Study IDs: B076201421922
Record Dates: First submitted 2018-06-19; First posted 2018-07-18 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: HIV Infections; Yellow Fever Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — sera or plasma samples to measure neutralizing antibodies against yellow fever
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HIV-infected patients: HIV-infected patients vaccinated at least once in their life against yellow fever
  Interventions: Diagnostic Test: Yellow fever neutralizing antibodies measure

INTERVENTIONS:
Diagnostic Test: Yellow fever neutralizing antibodies measure — Yellow fever neutralizing antibodies measure before vaccination, within the year after vaccination and at any delay after vaccination

SUMMARY:
Participating countries: Belgium

Context:

In June 2013, WHO notified that "a single dose of YF vaccine is sufficient to confer sustained life-long protective immunity against YF disease and that a booster dose is not necessary". . For HIV infected persons the recommendation was less stringent and the position paper concluded that hiv infected persons may "hypothetically, benefit from a second dose or booster dose ".1 Recently, WHO changed the recommendations about a booster dose of YF vaccine, based on the fact that serum neutralizing antibodies against YF are still at detectable levels after 20-35 years and probably lifelong in immunocompetent patients.

Unfortunately, data on persistence of Neutralizing antibodies Titers (NT) in immunocompromised patients are missing and only few studies reported data about HIV-infected patients. Additional data are needed.

Primary objective:

To assess presence / persistence of Neutralizing Titers (NT) of antibodies after YF immunization in HIV-infected patients.

Secondary objectives:

1. To identify risk factors for early and late waning of NT after YF immunization
2. To modelize kinetics of NT after YF immunization in different subpopulations of HIV patients, including population of young HIV patients infected vertically
3. To identify risk factors for absence of seroconversion in the year after YF immunization
4. To compare persistence of NT in HIV patients infected vertically or not vertically
5. To quantify seroconversion rate after YF vaccination Methodology / study design This study is a single arm, non randomized, cross-sectional, multicenter study in AIDS Reference Centers from Belgium.

The maximum duration of the study for each patient will be 1 visit, consisting of:

* the screening and inclusion visit (single visit V1) to check the patient eligibility, sign informed consent, perform the biologic tests necessary for the study and answer the questionnaire
* whenever possible, an additional serum / plasma sample coming from serabank / plasmabank will be identified for each patient. This sample must have been taken during the year following YF immunization.
* data about patient's HIV history has to be extracted from the HIV database or from patients' file

Estimated enrolment 750 patients + 30 patients infected vertically with HIV Primary outcome Number of HIV patients with protective YF NT ≥ 1:10 at different timepoints after YF immunization Secondary outcomes

1. Number of patients with protective YF NT ≥ 1:10 in the year following YF immunization
2. Risk factors (demographics and immunovirological parameters, antiretroviral treatment) for absence of seroconversion in the year following YF immunization
3. Risk factors (demographics and immunovirological parameters, antiretroviral treatment) of early waning (before 10 years) of YF NT
4. Risk factors (demographics and immunovirological parameters, antiretroviral treatment) of late waning (after 10 years) of YF NT Eligibility Inclusion criteria

1. Infection with HIV-1 (vertical transmission or not) 2. Immunization with at least one injection of YF vaccine (Stamaril®,17D strain Rockefeller, Sanofi Pasteur) with proof of vaccine administration 3. Informed consent signed prior to any study procedure Exclusion criteria Inability to give informed consent

Substudies

* Whenever possible, an additional sera or plasma sample from the year following YF vaccine will be selected and analyzed to assess early seroconversion rate
* Whenever possible, an additional sera or plasma sample from the year before YF vaccine will be selected and analyzed to assess seroconversion rate
* In CHU Saint-Pierre, an additional cohort of patients infected vertically with HIV will be selected and will participate to the study

DETAILED DESCRIPTION:
This study is a multicenter and cross sectional study performed in several ARC (AIDS Reference Centers) in Belgium and coordinated by CHU Saint-Pierre (Brussels, Belgium).

There is two parts in the study: a prospective part and a retrospective part. There is no control group in this study. Prospective study Sera / plasma samples of HIV patients immunized with at least one injection of YF vaccine (Stamaril® ,17D strain Rockefeller, Sanofi Pasteur) will be collected prospectively during the patient's single Visit. Analysis of samples will assess persistence of neutralizing antibodies titers (NT) against YF.

Retrospective study Whenever possible, serum or plasma sample will also be collected retrospectively (from a serum/plasma bank). Retrospective collection of samples must identify at least one sample per patient taken during the year before YF vaccine and from 30 days to 12 months following YF immunization

The retrospective study has three study timepoints :

Baseline is defined as an available sample during the period 12 months to day 0 before YF vaccination. Timepoint one is defined as a sample between one month and one year after YF.

In case of several samples, the sample nearest to one month will be chosen. Time point two is defined as the last available sample. In case the patient would have been re-vaccinated in the meantime (eg for interval higher than ten years; identied as DateVaccine2), the last sample before revaccination will be chosen.

Objectives of the retrospective study

1. To assess seroconversion rate during the year following YF immunization
2. To identify risk factors (demographics and immunovirological parameters, antiretroviral treatment ) for not seroconverting after primary vaccination with YF vaccine Description of the retrospective study Blood samples from HIV patients are kept, often for several years, in a sample bank. Depending of YF date of immunization, samples from the year before and following YF immunization will be identified and analysed. The PRNT technique will be used to assess presence of YF neutralizing antibodies (Serum or Plasma).

Samples will be centralized in CHU Saint-Pierre after one and two years of study. Assessment of presence of neutralizing antibodies titers (NT) against YF will be performed by PRNT (Plaque Reduction Neutralizing Test), which is the current gold standard technique.

After, the samples will be sent to France (Laboratory Cerba, Saint-Ouen l'Aumône) or in Germany (Berlin) to be analyzed. The surplus of your samples will be destroyed once the analyses described in this document have been carried out, i.e. in principle in maximum 10 years.

At least one sample will be analysed for each patient. A NT ≥ 1:10 will be considered as protective against natural YF.

Data that will be collected include demographics, date of HIV diagnosis, nadir CD4 and date, % CD4, CD38/CD8 (if available), CD4 and CD8 count at time of immunization against YF and at time of serological analysis, ARV therapy at time of immunization against YF and at time of serological analysis, plasma HIV RNA at time of immunization against YF and at time of serological analysis, number of YF vaccines, number of months with potential exposure to YF. Data will be collected by questionnaire and collected by local investigator, for instance by extraction from an HIV database. A CRF will then be completed by local investigators and sent to the data manager in CHU Saint-Pierre.

Vertical transmission substudy The same design is applied to this substudy. The population study is a population of HIV patients infected vertically, selected in only CHU Saint-Pierre.

Laboratory techniques:

Serological analysis will be performed at Centre for Biological Threats and Special Pathogens in Berlin, using a plaque reduction neutralization test (PRNT). This technique measures the neutralizing titers (NT: the highest serum dilution able to induce an 80% plaque reduction in cells infected by the YF17D strain). An YF virus NT ≥ 1:10 is accepted as a serologic surrogate marker of clinical protection against natural Yellow Fever.

Sampling and data collection:

Serological analysis will be performed on freezed sera/plasma samples (available from a serum/plasma bank retrospectively) or on fresh sera samples collected prospectively from HIV patients followed in different Belgian ARC. Samples will be centralized every year in CHU Saint-Pierre, Brussels.

Serological analysis will be performed at one timepoint for each patient after YF immunization to assess persistence of NT. When possible, it must also be performed on a freezed sample from the year before and following YF vaccine.

The following data will be collected, for instance extracted from HIV database of ARC: age, gender, mode of HIV contamination, ethnic origin, date of diagnosis of HIV, CD4 count nadir and date of nadir, history of AIDS, CD38/CD8 (if available), %CD4, CD4 and CD8 count, plasma HIV RNA at time of immunization against YF and at time of serological analysis, treatment for HIV at time of immunization against YF and at time of serological analysis, date of start of antiretroviral therapy.

Date(s) of YF immunization(s) will be checked with help of International Certificate of Immunization for Yellow Fever of every patient or with a medical note from Travel Clinic.

Potential natural YF exposure will be collected by patient questionnaire. All these data have to be included in the CRF completed by local investigator(s) then sent to the data manager in CHU Saint-Pierre.

The duration of the study for each patient is one single visit, consisting of the screening and inclusion visit (visit V1) to check the patient eligibility and to perform the biologic tests and exams necessary for the study.

ELIGIBILITY:
Inclusion Criteria:

* Infection with HIV-1 (vertically infected or not)
* Immunization with at least one injection of YF vaccine (Stamaril®,17D strain Rockefeller, Sanofi Pasteur) with proof of immunization
* Informed consent signed prior to any study procedure (for the Prospective part of the study )

Exclusion Criteria:

* Inability to give informed consent or incapacitation (for the Prospective part of the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SAMPLE SIZE Approximately 750 patients who meet the following inclusion criteria will be enrolled.
  Vertical transmission Substudy :
  Approximately 30 patients who meet the following inclusion criteria will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2023-01 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
Number of HIV patients with protective YF NT ≥ 1:10 at different timepoints after YF immunization | up to 60 years after YF vaccine administration
  protective YF NT ≥ 1:10

SECONDARY OUTCOMES:
Number of patients with protective YF NT ≥ 1:10 in the year following YF immunization | up to 1 year after YF immunization
  protective YF NT ≥ 1:10
Risk factors for absence of seroconversion in the year following YF immunization | up to 1 year after YF immunization
  Risk factors (demographics and immunovirological parameters, antiretroviral treatment, number of yellow fever vaccines)
Risk factors of early waning (before 10 years) of YF NT | before 10 years after YF immunization
  Risk factors (demographics and immunovirological parameters, antiretroviral treatment, number of YF vaccines)
Risk factors of late waning (after 10 years) of YF NT | after 10 years up to 60 years after YF vaccine administration
  Risk factors (demographics and immunovirological parameters, antiretroviral treatment, number of yellow fever vaccines)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Martin, MD, Principal Investigator — Centre Hospitalier Universitaire Saint Pierre
Locations (12):
- Belgium (12):
  - Instituut voor Tropische Geneeskunde, Antwerp
  - AZ Sint-Jan Brugge, Bruges
  - Centre Hospitalier Universitaire Saint-Pierre, Brussels
  - Hôpital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - CHU Charleroi Marie Curie, Charleroi
  - CHU Dinat Godinne, Dinant
  - UZ Gent, Ghent
  - Jessa Ziekenhuis, Hasselt
  - UZ Brussel, Jette
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège

IPD SHARING:
Plan to Share IPD: No